CLINICAL TRIAL: NCT03989830
Title: A Phase II Study of Second-line Chemotherapy Combined With Endostatin for Recurrent/Metastatic Head and Neck Epithelial Tumors That Cannot be Re-irradiated or Re-operated After Fist-line Platinum-based Chemotherapy
Brief Title: Second-Line Chemotherapy Combined With Endostatin for Recurrent/Metastatic HN Epithelial Tumors
Acronym: SLICER
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yan (Other)
Collaborators: Peking University (Other); Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor-Investigator, Sun Yan, MD, Professor, Chief of Head and Heck Group of Radiotherapy Department, Peking University Cancer Hospital, Peking University, Peking University
Organization: Peking University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJCH-2019YJZ24
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Head and Neck Neoplasms
Keywords: Endostatins; Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Drug Therapy; Endostatins; endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Second-line chemotherapy combined with Endostar (Experimental): Second-line chemotherapy+Endostar
  Interventions: Drug: second-line chemotherapy; Drug: Recombinant human endostatin

INTERVENTIONS:
Drug: second-line chemotherapy — choose appropriate regimen according to efficacy and adverse effects of first-line chemotherapy. q3W regimen, 6 cycles.
  Other Names: chemotherapy
Drug: Recombinant human endostatin — 7.5mg/m2/d，continuous intravenous pumping in 2ml/h for 5 days each cycle. Endostar(d-7) begins one week before chemotherapy(d0), first 5-day-pump(d-7 to d-2, 240ml, 2ml/h). Second 5-day-pump begins two days later (d1 to d5). the rest pumps can be done in the same manner. Three 5-day-pumps can be done during one chemotherapy cycle. Endostar will be pumped 18 weeks during 6 cycles'second-line chemotherapy.
  Other Names: Endostar

SUMMARY:
The prognoses of recurrent/metastatic head and neck epithelial tumors after first-line platinum-based chemotherapy is poor. The efficacy of second-line chemotherapy for those patients that cannot be re-irradiated or re-operated is limited according to NCCN guideline and other published data. This study was designed to evaluate the efficacy and safety of endostatin combined with second-line chemotherapy for patients of recurrent/metastatic head and neck epithelial tumors that cannot be re-irradiated or re-operated after fist-line platinum-based chemotherapy.

DETAILED DESCRIPTION:
The prognoses of recurrent/metastatic head and neck epithelial tumors after first-line platinum-based chemotherapy is poor. The efficacy of second-line chemotherapy for those patients that cannot be re-irradiated or re-operated is limited according to NCCN guideline and other published data. New agent for second-line treatment of recurrent and/or metastatic head and neck tumors is urgently needed. Recombinant human endostatin is an anti-angiogenetic target drug, which has been demonstrated a good efficacy for NSCLC. Studies about recombinant human endostatin in head and neck cancer mainly focus on NPC. And phase I study of endostatin combined with chemotherapy and/or radiotherapy for NPC showed a promising results.

This study was designed to evaluate the efficacy and safety of endostatin combined with second-line chemotherapy for patients of recurrent/metastatic head and neck epithelial tumors that cannot be re-irradiated or re-operated after fist-line platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old，<70 years old.
2. KPS ≥70.
3. Histopathology confirmed head and neck epithelial tumors, ie. Squamous cell carcinoma, adenocarcinoma, mucoepidermoid carcinoma, et al.
4. Relapse or metastasize after fist-line platinum-based chemotherapy，and the lesions cannot be re-irradiated or re-operated.
5. At least one measurable lesion (RECIST 1.1 version).
6. Life expectancy ≥ 6 months.
7. Adequate bone function: WBC≥3.0x109/L, ANC≥1.5 x109/L, HB≥90g/L, PLT≥100 x109/L. AST, ALT, Creatinine, urea nitrogen<1.25 ULN, normal coagulation function parameters.

Exclusion Criteria:

1. Malignant melanoma, lymphoma, other tumors from mesenchymal tissues.
2. Second primary malignant tumors.
3. Contraindications of chemotherapy: severe infections, significant cardiovascular disease, symptomatic arrythmia, uncontrolled diabetes mellitus, et al.
4. HIV infection, untreated chronic hepatitis B infection or carriers of HBV DNA copies >500IU/ml, active hepatitis C patients.
5. Uncontrolled hypertension.
6. Hemorrhagic tendency.
7. Epileptic seizure.
8. History of progression after anti-angiogenic target treatment.
9. History of allergy to recombinant human endostatin.
10. Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after the last dose of study treatment. Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment.
11. Receiving treatment of other clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2019-07-29 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | From the date of first drug administration, evaluation of response was performed every cycle during the treatment and then every 3 months after the completion of the treatment up to 36 months
  include complete remission, partial remission, and stable disease

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From the date of first drug administration, evaluation of response was performed every cycle during the treatment and then every 3 months after the completion of the treatment up to 36 months
  include complete remission and partial remission
Progress Free Survival (PFS) | From the date of first drug administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  1，2 years PFS
Overall Survival (OS) | From the date of first drug administration until the date of death, assessed up to 36 months
  1，2 years OS

CONTACTS AND LOCATIONS:
Overall Officials: Sun Yan, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The data is administered by Peking University Cancer Hospital, the investigators need to request related department for sharing IPD.

REFERENCES:
- [Background] Lu S, Li L, Luo Y, Zhang L, Wu G, Chen Z, Huang C, Guo S, Zhang Y, Song X, Yu Y, Zhou C, Li W, Liao M, Li B, Xu L, Chen P, Hu C, Hu C. A multicenter, open-label, randomized phase II controlled study of rh-endostatin (Endostar) in combination with chemotherapy in previously untreated extensive-stage small-cell lung cancer. J Thorac Oncol. 2015 Jan;10(1):206-11. doi: 10.1097/JTO.0000000000000343. PMID 25654728
- [Background] Cui C, Mao L, Chi Z, Si L, Sheng X, Kong Y, Li S, Lian B, Gu K, Tao M, Song X, Lin T, Ren X, Qin S, Guo J. A phase II, randomized, double-blind, placebo-controlled multicenter trial of Endostar in patients with metastatic melanoma. Mol Ther. 2013 Jul;21(7):1456-63. doi: 10.1038/mt.2013.79. Epub 2013 May 14. PMID 23670576
- [Background] Zhou J, Wang L, Xu X, Tu Y, Qin S, Yin Y. Antitumor activity of Endostar combined with radiation against human nasopharyngeal carcinoma in mouse xenograft models. Oncol Lett. 2012 Nov;4(5):976-980. doi: 10.3892/ol.2012.856. Epub 2012 Aug 8. PMID 23162635
- [Background] Wen QL, Meng MB, Yang B, Tu LL, Jia L, Zhou L, Xu Y, Lu Y. Endostar, a recombined humanized endostatin, enhances the radioresponse for human nasopharyngeal carcinoma and human lung adenocarcinoma xenografts in mice. Cancer Sci. 2009 Aug;100(8):1510-9. doi: 10.1111/j.1349-7006.2009.01193.x. Epub 2009 May 21. PMID 19459845
- [Background] Guan Y, Li A, Xiao W, Liu S, Chen B, Lu T, Zhao C, Han F. The efficacy and safety of Endostar combined with chemoradiotherapy for patients with advanced, locally recurrent nasopharyngeal carcinoma. Oncotarget. 2015 Oct 20;6(32):33926-34. doi: 10.18632/oncotarget.5271. PMID 26418895
- [Background] Jin T, Li B, Chen XZ. A phase II trial of Endostar combined with gemcitabine and cisplatin chemotherapy in patients with metastatic nasopharyngeal carcinoma (NCT01612286). Oncol Res. 2013;21(6):317-23. doi: 10.3727/096504014X13983417587401. PMID 25198661
- [Background] Ye W, Liu R, Pan C, Jiang W, Zhang L, Guan Z, Wu J, Ying X, Li L, Li S, Tan W, Zeng M, Kang T, Liu Q, Thomas GR, Huang M, Deng W, Huang W. Multicenter randomized phase 2 clinical trial of a recombinant human endostatin adenovirus in patients with advanced head and neck carcinoma. Mol Ther. 2014 Jun;22(6):1221-1229. doi: 10.1038/mt.2014.53. Epub 2014 Mar 25. PMID 24662947
- [Background] Hansma AH, Broxterman HJ, van der Horst I, Yuana Y, Boven E, Giaccone G, Pinedo HM, Hoekman K. Recombinant human endostatin administered as a 28-day continuous intravenous infusion, followed by daily subcutaneous injections: a phase I and pharmacokinetic study in patients with advanced cancer. Ann Oncol. 2005 Oct;16(10):1695-701. doi: 10.1093/annonc/mdi318. Epub 2005 Jul 12. PMID 16012180
- [Background] Li X, Gu G, Soliman F, Sanders AJ, Wang X, Liu C. The Evaluation of Durative Transfusion of Endostar Combined with Chemotherapy in Patients with Advanced Non-Small Cell Lung Cancer. Chemotherapy. 2018;63(4):214-219. doi: 10.1159/000493098. Epub 2018 Oct 22. PMID 30347389